CLINICAL TRIAL: NCT00745667
Title: The LAMA Trial: Laparoscopic Correction of Perforated Peptic Ulcer Versus Open Correction by Upper Laparotomy
Brief Title: The LAMA Trial: Laparoscopic Correction of Perforated Peptic Ulcer Versus Open Correction
Acronym: LAMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Gastrostart (Other)
Responsible Party: Drs. M.J.O.E. Bertleff, MD, Diaconessenhuis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAMA1; Gastrostart The Netherlands
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Perforated Peptic Ulcer
Keywords: laparoscopic; peptic ulcer
MeSH Terms: conditions — Peptic Ulcer Perforation; Peptic Ulcer | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): laparoscopic
  Interventions: Procedure: laparoscopic surgery
- 2 (Active Comparator): open correction
  Interventions: Procedure: Upper laparotomy

INTERVENTIONS:
Procedure: laparoscopic surgery — laparoscopic correction perforated peptic ulcer
  Arms: 1
Procedure: Upper laparotomy — upper laparotomy for correction of perforated peptic ulcer
  Arms: 2

SUMMARY:
This is a multicenter trial comparing laparoscopic correction of a perforated peptic ulcer with the open technique by upper laparotomy. Hypothesis is that after laparoscopic correction will be discharged 3 days sooner due to less postoperative pain and complications.

DETAILED DESCRIPTION:
as written above

ELIGIBILITY:
Inclusion Criteria:

* All patients clinical suspected for perforated peptic ulcer

Exclusion Criteria:

* Pregnancy
* Younger than 18 years
* Unable to sign consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 1999-07; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
days of discharge | 7 days

SECONDARY OUTCOMES:
postoperative VAs pain score and opiate usage; postoperative complications; Quality of live (RAND 36, euroquol) | follow up 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Johan Lange, PhD,MD, Study Director — Erasmus university hospital
Locations (1):
- Diaconessenhuis, Leiden, Netherlands